CLINICAL TRIAL: NCT06689930
Title: Dissemination and Implementation of a Community-driven Approach to Improve the Health of Women, Infants, and Families: Pre-implementation Phase to Adapt Staying Healthy After Childbirth (STAC)
Brief Title: Community-based Implementation of Adapted STAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1594; Protocol Approved 4/11/25 (Other: UW Madison); U48DP006793 (NIH)
Record Dates: First submitted 2024-11-07; First posted 2024-11-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Blood Pressure; Hypertension; Pregnancy Related; Health Equity
Keywords: Prenatal; Post Partum; Hypertensive Disorders of Pregnancy; Remote Patient Monitoring; Blood Pressure; Community-Based Participation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This is primarily a qualitative study designed to identify implementation strategies for the Adapted Staying Healthy After Childbirth (A-STAC). This pre-implementation phase includes 10 pilot participants and at least 2 CBO staff.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STAC-CAB Members (No Intervention): Staying Healthy After Childbirth - Community Advisory Board members (8-12 members)
- Lived Experience Group Members (No Intervention): Lived Experience Group members (8-12 members)
- PDSA Cycle Participants and CBO Staff (Experimental): Black pregnant or postpartum persons and Community Based Organization Staff
  Interventions: Other: PDSA Cycles

INTERVENTIONS:
Other: PDSA Cycles — Conduct PDSA cycle and follow-up interviews and surveys for patients (5 per cycle, 10 total) and CBO staff (no less than 2)
  Arms: PDSA Cycle Participants and CBO Staff

SUMMARY:
This study is being done to adapt the Staying Healthy After Childbirth (STAC) intervention for implementation among Black Women and Birthing Persons (WBP).

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy (HDP) are windows into chronic disease risk. The immediate postpartum (PP) period (6 weeks) is the highest risk and most important period for prevention of serious adverse outcomes with long term consequences. This project focuses on a multicomponent evidence-based intervention, Staying Healthy After Childbirth (STAC) that has been tested in a Midwest academic hospital. The intervention has been shown to be effective at addressing factors associated with health promotion priorities in populations with high levels of health disparities and inequities by increasing access to hypertension (HTN) care in the critical PP window by providing patients a home blood pressure monitor and access to a dedicated healthcare team that provides remote BP surveillance and antihypertensive medication titration. To optimize STAC to prevent and reduce racial disparities in immediate PP morbidity and mortality, deeper engagement with community stakeholders is critical.

This is a qualitative investigation designed as pre-implementation of the Adapted Staying Healthy After Childbirth (A-STAC) intervention.

STAC-Community Advisory Board (CAB) members and Lived Experience Group members will provide qualitative data through semi-structured interviews regarding implementation factors of STAC, including priorities for adaptation, barriers and facilitators to implementation, and usability. Rapid qualitative analysis will be used to glean themes from the qualitative data. A second round of semi-structured focus groups using the nominal decision-making process will be conducted to address the revisions to implementation strategies and determine priorities for A-STAC. Next, abbreviated study cycles to test implementation (Plan-Do-Study-Act or PDSA cycles) will take place, with a Community Based Organization (CBO) partner and participating Black pregnant persons. After each PDSA cycle, interviews and surveys with patients and staff will be conducted. Rapid qualitative analysis will again be used to gain information about the usability of A-STAC from the focus group; this information will then be used to refine the A-STAC intervention. This process will be repeated for a second PDSA cycle, after which the A-STAC intervention will be finalized for implementation (registered to a separate ClinicalTrials.gov record).

Step 1: Conduct interviews with STAC-CAB members (8-12 members) and Lived Experience Group members (8-12 members) to evaluate implementation factors and priorities for adaptation of STAC.

Use rapid qualitative analysis process to glean implementation strategies.

Step 2: Conduct small focus groups (3-4 participants per group) with STAC-CAB members (8-12 members) and Lived Experience Group members separately using nominal group decision decision making process.

Address revisions to implementation strategies and priorities for A-STAC.

Step 3: Conduct PDSA cycle and follow-up interviews and surveys for patients (5 participants per cycle, 10 total) and CBO staff (at least 2 staff).

Step 4: Incorporate usability data from cycle 1 to refine A-STAC.

Repeat steps 3-4 for second PDSA cycle.

Step 5: Finalize A-STAC Intervention.

ELIGIBILITY:
Inclusion Criteria (Interviews and Focus Groups):

* Belong to the STAC-CAB or Lived Experience Group
* Aged 18 or older

Inclusion Criteria (CBO Staff):

* Staff of CBO participating in PDSA cycle
* Aged 18 years or older

Inclusion Criteria (PDSA-Cycles):

* Pregnant persons greater than or equal to 24 weeks gestation and prior to delivery or postpartum
* Self-Identify as African American or Black
* Aged 18 years or older
* Capable of providing informed consent in English
* Can follow M•care System use instructions in English
* Have ownership of a functioning and reliable smartphone to upload and use the M•other App
* Interested in preventing or managing blood pressure during pregnancy

Exclusion Criteria (PDSA-Cycles):

* Persistent second or third trimester bleeding at time of enrollment
* Premature rupture of membranes in the current pregnancy at time of enrollment
* Known unrepaired maternal congenital heart disease requiring surgical correction
* Maternal heart failure
* Chronic kidney disease specifically requiring dialysis
* On greater than two antihypertensive medications at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Qualitative Summary of Barriers to Implementation of A-STAC | up to 4 weeks
  Barriers to implementation of A-STAC in CBOs will be investigated via qualitative analysis of interviews and focus groups with STAC-CAB members. All feedback regarding barriers will be coded for themes summarized by participant count.
Qualitative Summary of Facilitators to Implementation of A-STAC | up to 4 weeks
  Facilitators to implementation of A-STAC in CBOs will be investigated via qualitative analysis of interviews and focus groups with STAC-CAB members. All feedback regarding facilitators will be coded for themes summarized by participant count.
Qualitative Summary of Adaptations to STAC | up to 8 weeks
  Adaptations to STAC will be analyzed from patient participant interviews and CBO staff participants post-PDSA cycles. Interviews will be coded for themes summarized by count.
The Acceptability of Intervention Measure (AIM) | up to 8 weeks
  The Acceptability of Intervention Measure (AIM) measures intervention acceptability with 4 items ranked on a 5-point Likert-type scale from 1 = Completely Disagree to 5 = Completely Agree. Higher scores indicate higher acceptability.
The Intervention Appropriateness Measure (IAM) | up to 8 weeks
  The Intervention Appropriateness Measure (IAM) measures intervention appropriateness with 4 items ranked on a 5-point Likert-type scale from 1 = Completely Disagree to 5 = Completely Agree. Higher scores indicate higher acceptability.
The Feasibility of Intervention Measure (FIM) | up to 8 weeks
  The Feasibility of Intervention Measure (FIM) measures intervention feasibility with 4 items ranked on a 5-point Likert-type scale from 1 = Completely Disagree to 5 = Completely Agree. Higher scores indicate higher acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Hoppe, DO, PhD, Principal Investigator — University of Wisconsin, Madison; Andrew Garbacz, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: STAC Web Page — https://www.obgyn.wisc.edu/stac